CLINICAL TRIAL: NCT04758832
Title: The Effect of Poorly Designed School Furniture on Children's Head and Scapulae Postures: A Cross Sectional Design
Brief Title: The Effect of Poorly Designed School Furniture on Children's Head and Scapulae Postures
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Assistant. Professor of physical therapy, Department of Physical Therapy for Pediatrics, Delta University for Science and Technology
Other Study IDs: P.T.REC/012/003029
Record Dates: First submitted 2021-02-06; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Ergonomics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
investigate the compatibility of school furniture design

ELIGIBILITY:
Inclusion Criteria:

* had normal body mass index (ranged from 18.5 to 24.9 kg/ m2),
* The school furniture workstations used by all subjects were all of wooden flat desks and benches.

Exclusion Criteria:

* suffering from respiratory or heart problems

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Two hundred and fifty-seven normal children were evaluated for eligibility; thirty-five children were excluded because they failed to fulfill the inclusion criteria and sixteen parents refused to enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
weight | up to 24 weeks
  measured in kilograms
height | up to 24 weeks
  measured in centimetres
Body mass index (BMI) | up to 24 weeks
  It was calculated as the ratio of the subject's height (in meter) and weight (in kilogram) i.e. BMI= Weight/ Height2
anthropometric measurement for child | up to 24 weeks
  The anthropometric measurement for child were measured in mm by Auto CAD analysis for recorded photographs from sitting position.it include:1) elbow seat height: Measured with the elbow flexed at 90°, as the vertical distance from the bottom of the tip of the elbow to the student's seated surface, 2) shoulder height: Measured as the vertical distance from the top of the shoulder at the acromion process to the student's sitting surface,3) upper limb length: Difference between the elbow height and shoulder height.
anthropometric measurement for school furniture | up to 24 weeks
  The furniture dimensions were measured in mm by Auto CAD analysis for recorded photographs from sitting position.it include: 1) seat height: Measured as a distance from the floor to the highest point on the front of the seat, 2) seat depth: Measured from the back of the sitting surface of the seat to its front,3) backrest height: The vertical distance from the desk seat to the top edge of backrest, 4)desk- seat height: The vertical distance from the seat to the top of the front edge of the desk and 5) under surface of desk height: The vertical distance from the floor to the bottom of the front edge of the shelf under the writing surface..

SECONDARY OUTCOMES:
Correlation between educational furniture dimensions and the user body dimensions | through study completion, an average of 1 year.
  the percentage of compatibility for the ergonomics design of school furniture were tested by using the following equations: Equation (1): Seat height to popliteal height (N +2) cos 30°≤ SH < (N + 2) cos 5° Where SH is seat height and N is popliteal height). Equation (2): Seat depth to the popliteal-buttock length 80%M≤ SD < 95%M Where SD is seat depth and M is popliteal-buttock length. Equation (3): Backrest height:60% H≤ BH < 80% H Where BH is backrest height and H is shoulder height (scapula height). the previous equations represent the correlation between arthopemeteric measurements for the child (the user) and anthropometric measurement for school furniture.The percentage of matching and dis-matching school furniture calculated.
Head postures (angles) | through study completion, an average of 1 year.
  Auto CAD program (version 2013) used to determine head postures (angles). 1) Head flexion angle: Line of canthus to tragus with respect to vertical (measured from vertical above intersect). 2) Neck flexion angle : Line of tragus to C7 with respect to vertical (measured from vertical above intersect)
scapular postures (displacement and elevation). | through study completion, an average of 1 year.
  Auto CAD program (version 2013) used to determine scapular postures (displacement and elevation in mm). 1) Scapula displacement: Horizontal distance between markers at C7 and the anterior border of the acromion (measured in mm), 2)Scapula elevation: Vertical distance between markers at C7 and the anterior border of the acromion.

CONTACTS AND LOCATIONS:
Locations (1):
- AAA, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
will be shared at December 2021
Supporting Information: SAP, ICF